CLINICAL TRIAL: NCT06894784
Title: Semaglutide And Empagliflozin Combination Therapy Added To Automated Insulin Delivery In Adults With Type 1 Diabetes (SEMPA)
Brief Title: A Clinical Trial to Evaluate The Effects of Semaglutide and Empagliflozin Combined to Automated Insulin Delivery on Diabetes Control in Adults Living With Type 1 Diabetes
Acronym: SEMPA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Diabetes Canada (Other)
Responsible Party: Principal Investigator, Michael Tsoukas, Assistant Professor of Medicine, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-10723
Record Dates: First submitted 2025-03-07; First posted 2025-03-25 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Type 1
Keywords: T1D; Combination Therapy; Automated Insulin Delivery; SGLT2-i; GLP1-RA; Insulin; Artificial Pancreas; GLP-1 receptor agonist; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: 2×2 factorial, randomized, placebo-controlled, double-blind, crossover trial assessing the effects of Semaglutide and Empagliflozin, individually and combined, added to AID therapy.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide, Ozempic® (at maximum tolerated dose) + Automated Insulin Delivery system (Experimental): Semaglutide is a Glucagon-Like Peptide 1 Receptor Agonist. It stimulates GLP1 in the body, which allows for increased satiety, reduced glucagon levels, delayed gastric emptying, and in some, increased insulin secretion. It is a once per week subcutaneous injection.
  Participants will self-administer the colourless solution subcutaneously in the abdomen, thighs, or upper arms once weekly per the dosing schedule below.
  Weeks 1-4 : 0.25 mg (0.19 mL) Weeks 5-8 : 0.50 mg (0.38 mL) Weeks 9-12 : 1.0 mg (0.74 mL) Weeks 13-22 : 1.0 mg (0.74 mL)
  To match the recommendation from the product monograph and to ensure a steady state is reached before initiating the evaluation period, study drugs will be titrated for 12 weeks.
  Interventions: Drug: Intervention Period 1: Semaglutide + Empagliflozin; Drug: Intervention Period 2: Semaglutide + Empagliflozin Placebo; Drug: Intervention Period 3: Semaglutide Placebo + Empagliflozin; Drug: Intervention Period 4: Semaglutide Placebo + Empagliflozin Placebo
- Placebo + Automated Insulin Delivery system (Active Comparator): Participants will self-administer the colourless solution subcutaneously in the abdomen, thighs, or upper arms once weekly per the dosing schedule below.
  Weeks 1-4 : 0.19 mL Weeks 5-8 : 0.38 mL Weeks 9-12 : 0.74 mL Weeks 13-22 : 0.74 mL
  To match the recommendation from the product monograph and to ensure a steady state is reached before initiating the evaluation period, study drugs will be titrated for 12 weeks.
  Interventions: Drug: Intervention Period 1: Semaglutide + Empagliflozin; Drug: Intervention Period 2: Semaglutide + Empagliflozin Placebo; Drug: Intervention Period 3: Semaglutide Placebo + Empagliflozin; Drug: Intervention Period 4: Semaglutide Placebo + Empagliflozin Placebo

INTERVENTIONS:
Drug: Intervention Period 1: Semaglutide + Empagliflozin — Semaglutide Injection: Subcutaneous injection, titrated over 12 weeks to a stable dose (1 mg), administered weekly.
  Empagliflozin Tablet: Oral tablet (2.5 mg), administered daily.
  Automated Insulin Delivery (AID) System: Continuous use of the participant's personal commercial AID system.
Drug: Intervention Period 2: Semaglutide + Empagliflozin Placebo — Semaglutide Injection: Subcutaneous injection, titrated over 12 weeks to a stable dose (1 mg), administered weekly.
  Empagliflozin Placebo Tablet: Oral placebo tablet, matched in appearance to empagliflozin (2.5 mg), administered daily.
  Automated Insulin Delivery (AID) System: Continuous use of the participant's personal commercial AID system.
Drug: Intervention Period 3: Semaglutide Placebo + Empagliflozin — Semaglutide Placebo Injection: Subcutaneous placebo injection (titrated over 12 weeks to a stable 1 mg dose), matched in appearance to semaglutide, administered weekly.
  Empagliflozin Tablet: Oral tablet (2.5 mg), administered daily.
  Automated Insulin Delivery (AID) System: Continuous use of the participant's personal commercial AID system.
Drug: Intervention Period 4: Semaglutide Placebo + Empagliflozin Placebo — Semaglutide Placebo Injection: Subcutaneous placebo injection (titrated over 12 weeks to a stable 1 mg dose), matched in appearance to semaglutide, administered weekly.
  Empagliflozin Placebo Tablet: Oral placebo tablet (2.5 mg), matched in appearance to empagliflozin, administered daily.
  Automated Insulin Delivery (AID) System: Continuous use of the participant's personal commercial AID system.

SUMMARY:
The goal of this clinical trial is to learn if Empagliflozin and Semaglutide, individually and combined, added to Automated Insulin Delivery (AID) works to improve time-in-range in adults living with Type 1 Diabetes. It will also evaluate the safety of Empagliflozin and Semaglutide in this context.

The primary hypothesis of this study is :

- The combination therapy of semaglutide and empagliflozin will increase time-in-range compared to placebo when added to AID therapy.

The secondary hypotheses are :

* The combination therapy of semaglutide and empagliflozin will increase time-in-range compared to semaglutide alone when added to AID therapy.
* The combination of semaglutide and empagliflozin will increase time-in-range compared to empagliflozin alone when added to AID therapy.

In this study, the research team will compare Empagliflozin and Semaglutide to a placebo (a look-alike substance that contains no drug) to see if they improve time-in-range.

This study has four groups:

Group 1: semaglutide injection + empagliflozin tablet. Group 2: semaglutide injection + placebo tablet. Group 3: placebo injection + empagliflozin tablet. Group 4: placebo injection + placebo tablet.

This is a 2x2 factorial crossover study. This means that all participants will undergo both injection intervention (placebo and semaglutide) arms. Within each injection arm, participants will take both tablets (placebo and empagliflozin). By the end of the study, every participant will have taken part in each study group.

DETAILED DESCRIPTION:
This study is designed as a 2x2 factorial, randomized, placebo-controlled, double-blind, crossover trial to investigate the effects of semaglutide and empagliflozin, individually and combined, on time-in-range (TIR) in adults with type 1 diabetes (T1D) using automated insulin delivery (AID) systems.

1. Study Design and Randomization:

   Factorial Design: The 2x2 factorial design allows for the simultaneous assessment of two interventions (semaglutide and empagliflozin) and their interaction. This design efficiently explores the individual and combined effects of the drugs. Randomization: Participants will be randomized in a 1:1 ratio to determine the order of the semaglutide and placebo injections (Arm A: semaglutide first, Arm B: placebo first). Within each arm, the order of empagliflozin and placebo tablets will also be randomized 1:1. This ensures that any potential carryover effects are minimized. Double-Blind: Both participants and investigators will be blinded to the treatment assignments, minimizing bias in data collection and analysis. Crossover Design: Each participant will receive all four treatment combinations (semaglutide + empagliflozin, semaglutide + placebo, placebo + empagliflozin, placebo + placebo), allowing for within-subject comparisons and reducing inter-individual variability.
2. Study Procedures:

   Screening and Baseline: Participants will undergo a screening visit to confirm eligibility criteria. Baseline characteristics, including demographic data, medical history, and current diabetes management, will be collected. Titration Period (Semaglutide): A 12-week titration period for semaglutide will be implemented to achieve a stable dose and minimize gastrointestinal side effects. This gradual dose escalation will follow standard clinical practice. Intervention Periods (Four Weeks Each): Each participant will undergo four four-week intervention periods, representing the four treatment combinations. During each intervention period, participants will continue to use their AID system.

   Participants will receive daily injections (semaglutide or placebo) and daily tablets (empagliflozin or placebo) according to the randomization schedule. Washout Periods: A two to four-week washout period will be implemented between the semaglutide/placebo arms to eliminate any carryover effects of semaglutide. A one to seven-day washout period will be implemented between the empagliflozin/placebo tablet administrations. This short period is considered sufficient for the elimination of empagliflozin. CGM Data Collection:

   Continuous glucose monitoring (CGM) data will be collected throughout the study, with a focus on the four-week intervention periods. CGM data will be used to calculate the primary outcome (TIR) and secondary outcomes. Questionnaires: At the end of each four-week intervention period, participants will complete questionnaires to assess: Diabetes distress and treatment satisfaction. Adverse Event Monitoring: Adverse events will be recorded throughout the study, from informed consent to the end of participation.
3. Statistical Analysis:

   Intention-to-Treat (ITT) Analysis: Statistical analyses will be performed on an ITT basis, including all participants who were randomized. Factorial Analysis: The factorial design allows for the assessment of the main effects of semaglutide and empagliflozin, as well as their interaction. Mixed-Effects Models: Mixed-effects models will be used to account for repeated measures and within-subject variability. Descriptive Statistics: Descriptive statistics will be used to summarize baseline characteristics and outcome measures. Adverse Event Analysis: Adverse events will be summarized and analyzed for frequency and severity.
4. Safety Considerations:

Participants will be closely monitored for adverse events. Rescue medications will be available for hypoglycemic events. Participants will receive education on the safe use of semaglutide, empagliflozin, and the AID system. The investigators will have the right to remove any participant from the study at any time if they feel it is in the best interest of the participant.

ELIGIBILITY:
The inclusion criteria at the time of enrollment are:

* Males and females aged 18 or older.
* Clinical diagnosis of T1D for at least one year.
* Use of AID system for at least three months.
* Body Mass Index (BMI) ≥ 23 kg/m2.

The exclusion criteria are:

* Use of GLP1-RA within one month of admission.
* Use of SGLT2i within two weeks of admission.
* Planned or ongoing pregnancy.
* Breastfeeding.
* Severe hypoglycemic episode within three months of admission (defined as an event where blood glucose levels were < 4.0 mmol/L, resulting in seizure, loss of consciousness, or the need to present to the emergency department).
* Diabetic ketoacidosis episode within six months of admission.
* History of acute pancreatitis, chronic pancreatitis, or gallbladder disease.
* Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia type 2.
* Severe impairment of renal function with an eGFR < 30 mL/min/1.73 m2 within four months of admission. eGFR will be computed using the CKD-EPI method.
* Clinically significant diabetic retinopathy or gastroparesis, as per the investigator's judgement.
* Bariatric surgery within six months of admission.
* A serious medical or psychiatric illness that would likely interfere with participation in this study, as per the investigator's judgement.
* Inability or unwillingness to comply with safe diabetes management practices, as per the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Time-in-Range | At days 7, 35, 63 of the titration period and days 3 and 7 of each intervention.
  The percentage of time spent in target glucose range (3.9-10.0 mmol/L), between Semaglutide and Empagliflozin versus placebo, added to AID therapy.

SECONDARY OUTCOMES:
Overall Time In Range | At days 7, 35, 63 of the titration period and days 3 and 7 of each intervention.
  Percentage of time (%) spent in ranges of glucose levels : between 3.9 to 10 mmol/L
  Nota Bene: Secondary endpoints will be computed for (i) semaglutide and empagliflozin versus placebo, (ii) semaglutide and empagliflozin versus empagliflozin alone, (iii) semaglutide and empagliflozin versus semaglutide alone.
Optimal Time In Range | At days 7, 35, 63 of the titration period and days 3 and 7 of each intervention.
  Percentage of time (%) spent in ranges of glucose levels : between 3.9 to 7.8 mmol/L
  Nota Bene: Secondary endpoints will be computed for (i) semaglutide and empagliflozin versus placebo, (ii) semaglutide and empagliflozin versus empagliflozin alone, (iii) semaglutide and empagliflozin versus semaglutide alone.
Time In Hypoglycemia | At days 7, 35, 63 of the titration period and days 3 and 7 of each intervention.
  Percentage of time (%) spent in ranges of glucose levels : below 3.9 and 3.0 mmol/L
  Nota Bene: Secondary endpoints will be computed for (i) semaglutide and empagliflozin versus placebo, (ii) semaglutide and empagliflozin versus empagliflozin alone, (iii) semaglutide and empagliflozin versus semaglutide alone.
Time In Mild Hyperglycemia | At days 7, 35, 63 of the titration period and days 3 and 7 of each intervention.
  Percentage of time (%) spent in ranges of glucose levels : above 7.8 mmol/L
  Nota Bene: Secondary endpoints will be computed for (i) semaglutide and empagliflozin versus placebo, (ii) semaglutide and empagliflozin versus empagliflozin alone, (iii) semaglutide and empagliflozin versus semaglutide alone.
Time Above Range | At days 7, 35, 63 of the titration period and days 3 and 7 of each intervention.
  Percentage of time (%) spent in ranges of glucose levels : above 10 mmol/L
  Nota Bene: Secondary endpoints will be computed for (i) semaglutide and empagliflozin versus placebo, (ii) semaglutide and empagliflozin versus empagliflozin alone, (iii) semaglutide and empagliflozin versus semaglutide alone.
Time In Severe Hyperglycemia | At days 7, 35, 63 of the titration period and days 3 and 7 of each intervention.
  Percentage of time (%) spent in ranges of glucose levels : above 13.9 mmol/L
  Nota Bene: Secondary endpoints will be computed for (i) semaglutide and empagliflozin versus placebo, (ii) semaglutide and empagliflozin versus empagliflozin alone, (iii) semaglutide and empagliflozin versus semaglutide alone.
Total Insulin dose | At days 7, 35, 63 of the titration period and days 3 and 7 of each intervention.
  Total daily insulin dose (U/l)
  Nota Bene: Secondary endpoints will be computed for (i) semaglutide and empagliflozin versus placebo, (ii) semaglutide and empagliflozin versus empagliflozin alone, (iii) semaglutide and empagliflozin versus semaglutide alone.
Basal insulin dose | At days 7, 35, 63 of the titration period and days 3 and 7 of each intervention.
  Total daily basal dose (U/l)
  Nota Bene: Secondary endpoints will be computed for (i) semaglutide and empagliflozin versus placebo, (ii) semaglutide and empagliflozin versus empagliflozin alone, (iii) semaglutide and empagliflozin versus semaglutide alone.
Bolus insulin dose | At days 7, 35, 63 of the titration period and days 3 and 7 of each intervention.
  Total daily bolus dose (U/l)
  Nota Bene: Secondary endpoints will be computed for (i) semaglutide and empagliflozin versus placebo, (ii) semaglutide and empagliflozin versus empagliflozin alone, (iii) semaglutide and empagliflozin versus semaglutide alone.
Carbohydrate intake | At days 7, 35, 63 of the titration period and days 3 and 7 of each intervention.
  Average daily meal carbohydrate intake (grams/day)
  Nota Bene: Secondary endpoints will be computed for (i) semaglutide and empagliflozin versus placebo, (ii) semaglutide and empagliflozin versus empagliflozin alone, (iii) semaglutide and empagliflozin versus semaglutide alone.
Patient-reported outcomes | At the end of each intervention at weeks 16, 21, 29, 34
  Average scores (unit) of the questionnaire :
  - Diabetes Distress Scale
  Nota Bene: Secondary endpoints will be computed for (i) semaglutide and empagliflozin versus placebo, (ii) semaglutide and empagliflozin versus empagliflozin alone, (iii) semaglutide and empagliflozin versus semaglutide alone.
Patient-reported outcomes | At the end of each intervention at weeks 16, 21, 29, 34
  Average scores (unit) of the questionnaire:
  - Diabetes Treatment Satisfaction Questionnaire
  Nota Bene: Secondary endpoints will be computed for (i) semaglutide and empagliflozin versus placebo, (ii) semaglutide and empagliflozin versus empagliflozin alone, (iii) semaglutide and empagliflozin versus semaglutide alone.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Michael Tsoukas, Principal Investigator — Division of Endocrinology and Metabolism - McGill University Health Center; Dr. Melissa-Rosina Pasqua, Study Director — Division of Endocrinology and Metabolism - McGill University Health Center; Dr. Vanessa Tardio, Study Director — Division of Endocrinology and Metabolism - McGill University Health Center; Dr. Ahmad Haidar, Study Director — Department of Biomedical Engineering - McGill University
Locations (1):
- Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Protocol will be included upon finalization onto the website, as well as upon request.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Cohen E, Tsoukas MA, von Oettingen JE, Yale JF, Garfield N, Vallis M, et al. A Randomized Controlled Trial to Alleviate Carbohydrate Counting in Type 1 Diabetes with Automated Fiasp and Pramlintide Closed-Loop Delivery. New Orleans: American Diabetes Association Conference; 2022.
- [Background] Haidar A, Lovblom LE, Cardinez N, Gouchie-Provencher N, Orszag A, Tsoukas MA, Falappa CM, Jafar A, Ghanbari M, Eldelekli D, Rutkowski J, Yale JF, Perkins BA. Empagliflozin add-on therapy to closed-loop insulin delivery in type 1 diabetes: a 2 x 2 factorial randomized crossover trial. Nat Med. 2022 Jun;28(6):1269-1276. doi: 10.1038/s41591-022-01805-3. Epub 2022 May 12. PMID 35551290
- [Background] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185
- [Background] Bradley C. The diabetes treatment satisfaction questionnaire: DTSQ. Handbook of Psychology and Diabetes: a guide to psychological measurement in diabetes research and practice. 1994;111:132.
- [Background] Fisher L, Hessler D, Polonsky W, Strycker L, Masharani U, Peters A. Diabetes distress in adults with type 1 diabetes: Prevalence, incidence and change over time. J Diabetes Complications. 2016 Aug;30(6):1123-8. doi: 10.1016/j.jdiacomp.2016.03.032. Epub 2016 Apr 4. PMID 27118163
- [Background] Nordisk N. Ozempic® Product Monograph. 2017.
- [Background] Zinman B, Bhosekar V, Busch R, Holst I, Ludvik B, Thielke D, Thrasher J, Woo V, Philis-Tsimikas A. Semaglutide once weekly as add-on to SGLT-2 inhibitor therapy in type 2 diabetes (SUSTAIN 9): a randomised, placebo-controlled trial. Lancet Diabetes Endocrinol. 2019 May;7(5):356-367. doi: 10.1016/S2213-8587(19)30066-X. Epub 2019 Mar 1. PMID 30833170
- [Background] Eng C, Kramer CK, Zinman B, Retnakaran R. Glucagon-like peptide-1 receptor agonist and basal insulin combination treatment for the management of type 2 diabetes: a systematic review and meta-analysis. Lancet. 2014 Dec 20;384(9961):2228-34. doi: 10.1016/S0140-6736(14)61335-0. Epub 2014 Sep 11. PMID 25220191
- [Background] de Wit HM, Vervoort GM, Jansen HJ, de Grauw WJ, de Galan BE, Tack CJ. Liraglutide reverses pronounced insulin-associated weight gain, improves glycaemic control and decreases insulin dose in patients with type 2 diabetes: a 26 week, randomised clinical trial (ELEGANT). Diabetologia. 2014 Sep;57(9):1812-9. doi: 10.1007/s00125-014-3302-0. Epub 2014 Jun 20. PMID 24947583
- [Background] Fakhoury WK, Lereun C, Wright D. A meta-analysis of placebo-controlled clinical trials assessing the efficacy and safety of incretin-based medications in patients with type 2 diabetes. Pharmacology. 2010;86(1):44-57. doi: 10.1159/000314690. Epub 2010 Jul 12. PMID 20616619
- [Background] Du Q, Wang YJ, Yang S, Zhao YY, Han P. Liraglutide for the treatment of type 2 diabetes mellitus: a meta-analysis of randomized placebo-controlled trials. Adv Ther. 2014 Nov;31(11):1182-95. doi: 10.1007/s12325-014-0164-2. Epub 2014 Nov 12. PMID 25388240
- [Background] Dejgaard TF, Schmidt S, Frandsen CS, Vistisen D, Madsbad S, Andersen HU, Norgaard K. Liraglutide reduces hyperglycaemia and body weight in overweight, dysregulated insulin-pump-treated patients with type 1 diabetes: The Lira Pump trial-a randomized, double-blinded, placebo-controlled trial. Diabetes Obes Metab. 2020 Apr;22(4):492-500. doi: 10.1111/dom.13911. Epub 2019 Dec 19. PMID 31696598
- [Background] Ahren B, Hirsch IB, Pieber TR, Mathieu C, Gomez-Peralta F, Hansen TK, Philotheou A, Birch S, Christiansen E, Jensen TJ, Buse JB; ADJUNCT TWO Investigators. Efficacy and Safety of Liraglutide Added to Capped Insulin Treatment in Subjects With Type 1 Diabetes: The ADJUNCT TWO Randomized Trial. Diabetes Care. 2016 Oct;39(10):1693-701. doi: 10.2337/dc16-0690. Epub 2016 Aug 4. PMID 27493132
- [Background] Mathieu C, Zinman B, Hemmingsson JU, Woo V, Colman P, Christiansen E, Linder M, Bode B; ADJUNCT ONE Investigators. Efficacy and Safety of Liraglutide Added to Insulin Treatment in Type 1 Diabetes: The ADJUNCT ONE Treat-To-Target Randomized Trial. Diabetes Care. 2016 Oct;39(10):1702-10. doi: 10.2337/dc16-0691. Epub 2016 Aug 9. PMID 27506222
- [Background] Johansen NJ, Dejgaard TF, Lund A, Schluntz C, Frandsen CS, Forman JL, Wewer Albrechtsen NJ, Holst JJ, Pedersen-Bjergaard U, Madsbad S, Vilsboll T, Andersen HU, Knop FK. Efficacy and safety of meal-time administration of short-acting exenatide for glycaemic control in type 1 diabetes (MAG1C): a randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2020 Apr;8(4):313-324. doi: 10.1016/S2213-8587(20)30030-9. Epub 2020 Mar 2. PMID 32135138
- [Background] Ahmann AJ, Capehorn M, Charpentier G, Dotta F, Henkel E, Lingvay I, Holst AG, Annett MP, Aroda VR. Efficacy and Safety of Once-Weekly Semaglutide Versus Exenatide ER in Subjects With Type 2 Diabetes (SUSTAIN 3): A 56-Week, Open-Label, Randomized Clinical Trial. Diabetes Care. 2018 Feb;41(2):258-266. doi: 10.2337/dc17-0417. Epub 2017 Dec 15. PMID 29246950
- [Background] Pratley RE, Aroda VR, Lingvay I, Ludemann J, Andreassen C, Navarria A, Viljoen A; SUSTAIN 7 investigators. Semaglutide versus dulaglutide once weekly in patients with type 2 diabetes (SUSTAIN 7): a randomised, open-label, phase 3b trial. Lancet Diabetes Endocrinol. 2018 Apr;6(4):275-286. doi: 10.1016/S2213-8587(18)30024-X. Epub 2018 Feb 1. PMID 29397376
- [Background] Capehorn MS, Catarig AM, Furberg JK, Janez A, Price HC, Tadayon S, Verges B, Marre M. Efficacy and safety of once-weekly semaglutide 1.0mg vs once-daily liraglutide 1.2mg as add-on to 1-3 oral antidiabetic drugs in subjects with type 2 diabetes (SUSTAIN 10). Diabetes Metab. 2020 Apr;46(2):100-109. doi: 10.1016/j.diabet.2019.101117. Epub 2019 Sep 17. PMID 31539622
- [Background] Gerstein HC, Colhoun HM, Dagenais GR, Diaz R, Lakshmanan M, Pais P, Probstfield J, Riesmeyer JS, Riddle MC, Ryden L, Xavier D, Atisso CM, Dyal L, Hall S, Rao-Melacini P, Wong G, Avezum A, Basile J, Chung N, Conget I, Cushman WC, Franek E, Hancu N, Hanefeld M, Holt S, Jansky P, Keltai M, Lanas F, Leiter LA, Lopez-Jaramillo P, Cardona Munoz EG, Pirags V, Pogosova N, Raubenheimer PJ, Shaw JE, Sheu WH, Temelkova-Kurktschiev T; REWIND Investigators. Dulaglutide and cardiovascular outcomes in type 2 diabetes (REWIND): a double-blind, randomised placebo-controlled trial. Lancet. 2019 Jul 13;394(10193):121-130. doi: 10.1016/S0140-6736(19)31149-3. Epub 2019 Jun 9. PMID 31189511
- [Background] Mann JFE, Orsted DD, Brown-Frandsen K, Marso SP, Poulter NR, Rasmussen S, Tornoe K, Zinman B, Buse JB; LEADER Steering Committee and Investigators. Liraglutide and Renal Outcomes in Type 2 Diabetes. N Engl J Med. 2017 Aug 31;377(9):839-848. doi: 10.1056/NEJMoa1616011. PMID 28854085
- [Background] Greco EV, Russo G, Giandalia A, Viazzi F, Pontremoli R, De Cosmo S. GLP-1 Receptor Agonists and Kidney Protection. Medicina (Kaunas). 2019 May 31;55(6):233. doi: 10.3390/medicina55060233. PMID 31159279
- [Background] Marso SP, Bain SC, Consoli A, Eliaschewitz FG, Jodar E, Leiter LA, Lingvay I, Rosenstock J, Seufert J, Warren ML, Woo V, Hansen O, Holst AG, Pettersson J, Vilsboll T; SUSTAIN-6 Investigators. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2016 Nov 10;375(19):1834-1844. doi: 10.1056/NEJMoa1607141. Epub 2016 Sep 15. PMID 27633186
- [Background] Marso SP, Daniels GH, Brown-Frandsen K, Kristensen P, Mann JF, Nauck MA, Nissen SE, Pocock S, Poulter NR, Ravn LS, Steinberg WM, Stockner M, Zinman B, Bergenstal RM, Buse JB; LEADER Steering Committee; LEADER Trial Investigators. Liraglutide and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):311-22. doi: 10.1056/NEJMoa1603827. Epub 2016 Jun 13. PMID 27295427
- [Background] Kielgast U, Holst JJ, Madsbad S. Treatment of type 1 diabetic patients with glucagon-like peptide-1 (GLP-1) and GLP-1R agonists. Curr Diabetes Rev. 2009 Nov;5(4):266-75. doi: 10.2174/157339909789804413. PMID 19925391
- [Background] Nauck MA, Holst JJ, Willms B, Schmiegel W. Glucagon-like peptide 1 (GLP-1) as a new therapeutic approach for type 2-diabetes. Exp Clin Endocrinol Diabetes. 1997;105(4):187-95. doi: 10.1055/s-0029-1211750. PMID 9285204
- [Background] Kobayati A, Haidar A, Tsoukas MA. Glucagon-like peptide-1 receptor agonists as adjunctive treatment for type 1 diabetes: Renewed opportunities through tailored approaches? Diabetes Obes Metab. 2022 May;24(5):769-787. doi: 10.1111/dom.14637. Epub 2022 Mar 2. PMID 34989070
- [Background] Stonehouse AH, Darsow T, Maggs DG. Incretin-based therapies. J Diabetes. 2012 Mar;4(1):55-67. doi: 10.1111/j.1753-0407.2011.00143.x. PMID 21707956
- [Background] Muller TD, Finan B, Bloom SR, D'Alessio D, Drucker DJ, Flatt PR, Fritsche A, Gribble F, Grill HJ, Habener JF, Holst JJ, Langhans W, Meier JJ, Nauck MA, Perez-Tilve D, Pocai A, Reimann F, Sandoval DA, Schwartz TW, Seeley RJ, Stemmer K, Tang-Christensen M, Woods SC, DiMarchi RD, Tschop MH. Glucagon-like peptide 1 (GLP-1). Mol Metab. 2019 Dec;30:72-130. doi: 10.1016/j.molmet.2019.09.010. Epub 2019 Sep 30. PMID 31767182
- [Background] Ahren B. Glucagon-like peptide-1 (GLP-1): a gut hormone of potential interest in the treatment of diabetes. Bioessays. 1998 Aug;20(8):642-51. doi: 10.1002/(SICI)1521-1878(199808)20:83.0.CO;2-K. PMID 9780839
- [Background] Gutzwiller JP, Drewe J, Goke B, Schmidt H, Rohrer B, Lareida J, Beglinger C. Glucagon-like peptide-1 promotes satiety and reduces food intake in patients with diabetes mellitus type 2. Am J Physiol. 1999 May;276(5):R1541-4. doi: 10.1152/ajpregu.1999.276.5.R1541. PMID 10233049
- [Background] Pasqua MR, Jafar A, Kobayati A, Tsoukas MA, Haidar A. Low-Dose Empagliflozin as Adjunct to Hybrid Closed-Loop Insulin Therapy in Adults With Suboptimally Controlled Type 1 Diabetes: A Randomized Crossover Controlled Trial. Diabetes Care. 2023 Jan 1;46(1):165-172. doi: 10.2337/dc22-0490. PMID 36331522
- [Background] Haidar A, Yale JF, Lovblom LE, Cardinez N, Orszag A, Falappa CM, Gouchie-Provencher N, Tsoukas MA, El Fathi A, Rene J, Eldelekli D, Lanctot SO, Scarr D, Perkins BA. Reducing the need for carbohydrate counting in type 1 diabetes using closed-loop automated insulin delivery (artificial pancreas) and empagliflozin: A randomized, controlled, non-inferiority, crossover pilot trial. Diabetes Obes Metab. 2021 Jun;23(6):1272-1281. doi: 10.1111/dom.14335. Epub 2021 Feb 28. PMID 33528904
- [Background] Rosenstock J, Marquard J, Laffel LM, Neubacher D, Kaspers S, Cherney DZ, Zinman B, Skyler JS, George J, Soleymanlou N, Perkins BA. Empagliflozin as Adjunctive to Insulin Therapy in Type 1 Diabetes: The EASE Trials. Diabetes Care. 2018 Dec;41(12):2560-2569. doi: 10.2337/dc18-1749. Epub 2018 Oct 4. PMID 30287422
- [Background] Tsoukas MA, Woo V, Tobe SW, Slee A, Rapattoni W, Ang FG, Seufert J, Neuen BL, Arnott C, Mahaffey KW, Wheeler DC. Cardiovascular and kidney outcomes with canagliflozin according to type 2 diabetes treatment targets at baseline: Data from the CANVAS programme and CREDENCE. Diabetes Obes Metab. 2023 Jul;25(7):2038-2042. doi: 10.1111/dom.15057. Epub 2023 Apr 4. No abstract available. PMID 36942888
- [Background] Riddle MC, Cefalu WT. SGLT Inhibitors for Type 1 Diabetes: An Obvious Choice or Too Good to Be True? Diabetes Care. 2018 Dec;41(12):2444-2447. doi: 10.2337/dci18-0041. No abstract available. PMID 30459245
- [Background] Pradhan A, Vohra S, Vishwakarma P, Sethi R. Review on sodium-glucose cotransporter 2 inhibitor (SGLT2i) in diabetes mellitus and heart failure. J Family Med Prim Care. 2019 Jun;8(6):1855-1862. doi: 10.4103/jfmpc.jfmpc_232_19. PMID 31334145
- See also: Sizar O, Podder V, Talati R. Empagliflozin. In: StatPearls. StatPearls Publishing; 2024. Accessed April 15, 2024 — http://www.ncbi.nlm.nih.gov/books/NBK532925/
- See also: Ozempic® Side Effects | Ozempic® (semaglutide) injection. Accessed April 15, 2024 — https://www.ozempic.com/how-to-take/side-effects.html